CLINICAL TRIAL: NCT02538250
Title: Acceptability Study on Nutricomp Drink Plus in Adult Patients
Brief Title: Acceptability Study on Oral Nutrition Supplement (ONS)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: B. Braun Medical UK Ltd. (Industry)
Responsible Party: Sponsor
Organization: B. Braun Melsungen AG (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: HC-G-H-1422
Record Dates: First submitted 2015-06-24; First posted 2015-09-02 (Estimated); Last update posted 2016-10-13 (Estimated); Status verified 2016-10

CONDITIONS: Oral Nutritional Supplementation
Keywords: Oral nutritional supplement; supplementation; adult patients

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 Nutricomp Drink Plus (Experimental): Nutricomp Drink Plus
  Interventions: Dietary Supplement: Nutricomp Drink Plus

INTERVENTIONS:
Dietary Supplement: Nutricomp Drink Plus — Oral nutritional supplementation

SUMMARY:
Required for Advisory Committee for Borderline Substances (ACBS) approval. Aim of this study is to access the palatability, compliance and GI-tolerance of Nutricomp® Drink Plus to show that it is acceptable for patients in the United Kingdom.

ELIGIBILITY:
Inclusion:

* Male and female patients
* ≥ 18 years of age
* Patients of the intended target group (e.g. MUST score ≥ 1) with an anticipated period of nutritional support ≥ 7 days
* Patient is able and willing to provide written informed consent

Exclusion:

* Hypersensitivity to milk, whey, soy, fish or any of the active substances or excipients
* Patients with available or potential impairment of sense of taste or smell due to disease (e.g. patients with cold, cancer patients) or medication (e.g. D-Penicillamine)
* Patients who express general dislike to two or more of the four flavours
* Severely impaired gastrointestinal function or complete failure
* Severe metabolic or circulatory disorders
* Acute disease
* Unstable vital functions
* Necessity of total parenteral nutrition or more than 50% Parenteral Nutrition in combined therapy
* Simultaneous participation in another interventional study
* Patients who are unwilling or mentally and/or physically unable to adhere to study procedures
* Pregnancy
* Emergencies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2015-07; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Occurrence of gastrointestinal tolerance parameters (Diarrhoea, Constipation, Bloating, Distension, Nausea, Vomiting, Burping, Regurgitation, Flatulence, Abdominal discomfort, Abdominal pain, Other (further gastrointestinal adverse events) | 7 days
  Parameters asked as required for acceptability studies by Advisory Committee for Borderline Substances- documented in a patient diary

SECONDARY OUTCOMES:
Occurrence of further adverse effects | 7 days
Evaluation of palatability by questionnaire | 1 day
  Five point hedonic scale
Evaluation of compliance. | 7 days
  Comparison of prescription and actual intake

CONTACTS AND LOCATIONS:
Overall Officials: David Sanders, Prof., Principal Investigator — The Royal Hallamshire Hospital,Regional Gastrointestinal and Liver Unit, Sheffield, UK
Locations (1):
- Sheffield Teaching Hospitals NHS Foundation Trust, The Royal Hallamshire Hospital, Regional Gastrointestinal and Liver Unit, Sheffield, United Kingdom